CLINICAL TRIAL: NCT03158831
Title: Drug Challenges Without Prior Skin Testing
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Elina Jerschow, Associate Professor of Clinical Medicine, Montefiore Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015-5610
Record Dates: First submitted 2017-05-11; First posted 2017-05-18 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Drug Hypersensitivity; Penicillin Allergy; Antibiotic Allergy
Keywords: Drug Allergy; Penicillin Allergy; Antibiotic Allergy; Graded Drug Challenge
MeSH Terms: conditions — Drug Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Prospective interventional study whereby each eligible patient undergoes a placebo-controlled graded challenge. Each patient receives a placebo prior to undergoing a graded challenge to 1/10 the treatment dose of the challenge drug followed by a full treatment dose of the challenge drug.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Placebo-Controlled Graded Drug Challenge (Other): This is a single arm study. All patients will receive a placebo prior to a graded drug challenge. Each patient serves as his/her own control.
  Interventions: Drug: Placebo-Controlled Graded Drug Challenge

INTERVENTIONS:
Drug: Placebo-Controlled Graded Drug Challenge — All patients receive a placebo followed by 30 minutes of observation. Patients then receive 1/10 of the treatment dose of the challenge drug followed by 30 minutes of observation. If no reaction, they will then receive a full dose of their challenge drug followed by 1 hour of observation. If they do not experience any reactions, they are deemed not to be allergic. All patients are asked to monitor for delayed reactions after the challenge. Patients are also called within 1 month of the challenge to determine if any delayed reactions occurred. Patients are called again within 1 year of the challenge to determine if they have subsequently taken the challenge drug and experienced any reactions.

SUMMARY:
The investigators are conducting a prospective study to determine the safety and outcomes of placebo-controlled graded drug challenges without prior skin testing in patients with a low-risk history of antibiotic hypersensitivity reaction based on history alone. The investigators hypothesize that the rate of reaction to graded drug challenges without prior skin testing in patients with a low-risk history of drug hypersensitivity reaction based on history alone will not be meaningfully more than the rate of reaction to placebo. The investigators hypothesize that the rate of adverse reactions to drug challenges without prior skin testing will not be meaningfully more than the rate of adverse reactions with prior skin testing as was observed in the investigators' historical clinic cohort.

DETAILED DESCRIPTION:
Graded drug challenges are the gold standard to exclude an immediate hypersensitivity reaction in patients with a low likelihood of drug allergy and are considered standard of care. Patients who tolerate a graded challenge are deemed to not be allergic to the drug and are not at increased risk for future reactions compared with the general population. Prior studies of graded challenges in appropriately selected patients have demonstrated low reaction rates with symptoms that were mainly mild and subjective in nature. The investigators are conducting a prospective study to determine the safety and outcomes of placebo-controlled graded drug challenges without prior skin testing in patients with a low-risk history of antibiotic hypersensitivity reaction based on history alone. Skin testing requires a separate visit and is, therefore, more time-consuming and costly than performing a graded challenge without skin testing. The investigators believe that they can determine if patients are at low-risk to react to an antibiotic based on a detailed history and, therefore, do not require skin testing prior to a challenge. Given the majority of symptoms to graded drug challenges reported in prior studies were mild and subjective, the investigators hypothesize that the rate of reaction to graded drug challenges without prior skin testing in patients with a low-risk history of drug hypersensitivity reaction based on history alone will not be meaningfully more than the rate of reaction to placebo. The investigators hypothesize that the rate of adverse reactions to drug challenges without prior skin testing will be not meaningfully more than the rate of adverse reactions with prior skin testing as was observed in the investigators' historical clinic cohort. All patients age 7 years or older with a history of a non-life-threatening reaction to an antibiotic are eligible to participate in a placebo-controlled graded drug challenge. The challenge is comprised of placebo followed by 30 minutes of observation, 1/10th of the treatment dose of the antibiotic the patient reported a reaction followed by 30 minutes of observation, and the full dose of the antibiotic followed by 1 hour of observation. All patients will be contacted via telephone within one month of a negative challenge to determine whether they experienced a delayed reaction. All patients will also be contacted via telephone within one year of a negative challenge to determine if they have safely taken the challenge drug.

ELIGIBILITY:
Inclusion Criteria:

* All patients seven years of age or older who have a low-risk, non-life-threatening history of adverse reaction to an antibiotic.

Exclusion Criteria:

* Patients under the age of seven.
* Pregnant patients.
* Patients with a history of a drug reaction that is high-risk and life-threatening including life-threatening angioedema, bronchospasm, or anaphylactic shock or a history of severe non-IgE-mediated reactions including serum sickness, Stevens-Johnson syndrome, toxic epidermal necrolysis, interstitial nephritis, hepatitis, hemolytic anemia, DRESS, skin and/or oral blisters, hypersensitivity vasculitis, pneumonitis, or pulmonary fibrosis.
* Patients who have taken antihistamines within 3 days of the drug challenge.

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2016-01-13 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Rate of unexpected reaction to graded drug challenges without prior skin testing compared to rate of unexpected reaction to graded drug challenges with prior skin testing. | It is anticipated the study will take 2 years to enroll 200 patients with subsequent data comparison.
  Determine the rate of unexpected reaction to a graded drug challenge without prior skin testing versus the rate of reaction to a graded drug challenge with prior skin testing in the investigators' historical cohort (data on this cohort has already been published: Iammatteo M, Ferastraoaru D, Koransky R, Alvarez-Arango S, Thota N, Akenroye A, Jerschow E. Identifying Allergic Drug Reactions Through Placebo-Controlled Graded Challenges. J Allergy Clin Immunol Pract. 2017 May - Jun;5(3):711-717.e2.).

SECONDARY OUTCOMES:
Rate of unexpected reaction to graded drug challenges versus placebos | Patients are monitored for 1 hour after completion of their drug challenge.
  Determine the rate of unexpected reaction to graded drug challenges without prior skin tests versus the rate of unexpected reaction to placebos in patients with a low-risk history of drug hypersensitivity reaction based on history alone.
Rate of unexpected delayed reaction to graded drug challenges | Patients are called within 1 month of their challenge to determine if they had any delayed reactions.
  Determine the rate of unexpected delayed reaction to graded challenges

CONTACTS AND LOCATIONS:
Overall Officials: Elina Jerschow, MD, MSc, Principal Investigator — Montefiore Medical Center/Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to make IPD available to other researchers.

REFERENCES:
- [Background] Iammatteo M, Ferastraoaru D, Koransky R, Alvarez-Arango S, Thota N, Akenroye A, Jerschow E. Identifying Allergic Drug Reactions Through Placebo-Controlled Graded Challenges. J Allergy Clin Immunol Pract. 2017 May-Jun;5(3):711-717.e2. doi: 10.1016/j.jaip.2016.09.041. Epub 2016 Nov 23. PMID 27888028
- [Background] Iammatteo M, Blumenthal KG, Saff R, Long AA, Banerji A. Safety and outcomes of test doses for the evaluation of adverse drug reactions: a 5-year retrospective review. J Allergy Clin Immunol Pract. 2014 Nov-Dec;2(6):768-74. doi: 10.1016/j.jaip.2014.08.001. Epub 2014 Sep 10. PMID 25439369
- [Background] Macy E, Romano A, Khan D. Practical Management of Antibiotic Hypersensitivity in 2017. J Allergy Clin Immunol Pract. 2017 May-Jun;5(3):577-586. doi: 10.1016/j.jaip.2017.02.014. Epub 2017 Mar 29. PMID 28365277
- [Background] Joint Task Force on Practice Parameters; American Academy of Allergy, Asthma and Immunology; American College of Allergy, Asthma and Immunology; Joint Council of Allergy, Asthma and Immunology. Drug allergy: an updated practice parameter. Ann Allergy Asthma Immunol. 2010 Oct;105(4):259-273. doi: 10.1016/j.anai.2010.08.002. PMID 20934625